CLINICAL TRIAL: NCT01488682
Title: The Safety and Efficacy of the Harmonic Scalpel in Neck Dissection : A Prospective Randomized Study
Brief Title: The Safety and Efficacy of the Harmonic Scalpel in Neck Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2011-0014
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; Neck dissection; Harmonic scalpel
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Neck Dissection

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Harmonic scalpel (Experimental): Harmonic Focus® Curved Shears (Ethicon Endo-Surgery, Cincinnati, OH) was used for vascular control of the surgery regardless of vessel diameter, except when hand-tied or suture ligation was needed for IJV ligation or in case bleeding was not controlled with electrocoagulation
  Interventions: Procedure: Neck dissection with Harmonic scalpel
- conventional hand tie ligation (Active Comparator): electrocautery was used to control the small vessels and conventional hand-tied ligation was used for large sized arterial, venous, or lymphatic vessels.
  Interventions: Procedure: neck dissection with conventional hand-tie ligation

INTERVENTIONS:
Procedure: Neck dissection with Harmonic scalpel — The Harmonic Focus® Curved Shears (Ethicon Endo-Surgery, Cincinnati, OH) was used for vascular control of the surgery regardless of vessel diameter, except when hand-tied or suture ligation was needed for IJV ligation or in case bleeding was not controlled with electrocoagulation
  Other Names: Harmonic Focus® Curved Shears
  Arms: Harmonic scalpel
Procedure: neck dissection with conventional hand-tie ligation — electrocautery was used to control the small vessels and conventional hand-tied ligation was used for large sized arterial, venous, or lymphatic vessels
  Arms: conventional hand tie ligation

SUMMARY:
Recently, the HS has been used in head and neck surgery as an alternative to conventional hand-tied ligation for hemostasis, which is a time-consuming procedure. Limited data have been published on the evidence of its safety in ND, especially in radical ND. Researchers investigated the safety and efficacy of the Harmonic scalpel (HS) in neck dissection (ND), while using conventional hand-tied ligation to a minimum, in terms of operating time, blood loss, drainage and complications.

ELIGIBILITY:
Inclusion Criteria:

* preoperative diagnosis of head and neck squamous cell carcinoma
* surgery as initial treatment

Exclusion Criteria:

* cases in which the ND specimen could not be separated from the primary tumor
* past history of neck surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
number of harvested lymph nodes | when the pathologist examine the specimen which is within 1 week after operation
  number of harvested lymph nodes counted from the lymphfatty tissue after neck dissection
intra-operative surgery-related complications | complicated events will be monitored during the operation which takes 60 min to 160 min according to the extent of surgery
  major vessel laceration, major nerve injury, and penetration into adjacent vital structures such as trachea or esophagus
post-operative complications | participants will be followed for 1 month after the surgery
  hemorrhage, hematoma, seroma, chylous leakage, and neurologic complications

SECONDARY OUTCOMES:
operating time | when the neck dissection specimen is removed from the patient at an average time of 60 min to 160 min according to the extent of surgery
  The time from the first procedure after subplatysmal flap elevation to removal of neck dissection specimen will be measured
intraoperative bleeding | The amount will be estimated at the end of the surgery at an average time of 60 min to 160 min according to the extent of surgery
  Estimated blood loss from the collection bottle for the suction drain (ml) will be measured
total amount of drainage | estimated until the drain tube is removed at the average of 4 to 7 days according to the extent of surgery
  total amount of drainage is estimated from the collection bottle of closed drain(ml)
duration of drain placement | estimated at 6AM daily, until the drain is removed at an average of 4 to 7 days according to the extent of surgery
  amount of drain collected in the drain bottle is estimated daily (ml)
days of hospital stay | documented when the patient leaves the hospital at an average time of 10 to 28 days according to the extent of surgery
  duration of hospital stay by days

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] McCarus SD. Physiologic mechanism of the ultrasonically activated scalpel. J Am Assoc Gynecol Laparosc. 1996 Aug;3(4):601-8. doi: 10.1016/s1074-3804(05)80174-4. PMID 9050696
- [Result] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Result] BuSaba NY, Schaumberg DA. Predictors of prolonged length of stay after major elective head and neck surgery. Laryngoscope. 2007 Oct;117(10):1756-63. doi: 10.1097/MLG.0b013e3180de4d85. PMID 17690609
- [Result] Patel RS, McCluskey SA, Goldstein DP, Minkovich L, Irish JC, Brown DH, Gullane PJ, Lipa JE, Gilbert RW. Clinicopathologic and therapeutic risk factors for perioperative complications and prolonged hospital stay in free flap reconstruction of the head and neck. Head Neck. 2010 Oct;32(10):1345-53. doi: 10.1002/hed.21331. PMID 20091687
- [Result] Smith TL, Smith JM. Electrosurgery in otolaryngology-head and neck surgery: principles, advances, and complications. Laryngoscope. 2001 May;111(5):769-80. doi: 10.1097/00005537-200105000-00004. PMID 11359154
- [Result] Roth JH, Urbaniak JR, Boswick JM. Comparison of suture ligation, bipolar cauterization, and hemoclip ligation in the management of small branching vessels in a rat model. J Reconstr Microsurg. 1984 Jul;1(1):7-9. doi: 10.1055/s-2007-1007047. PMID 6544345
- [Result] Ellman BR. New instrument for rapid hemostasis and division of small vessels. Am J Surg. 1982 Jun;143(6):772-3. doi: 10.1016/0002-9610(82)90058-7. PMID 7091517
- [Result] Amaral JF. Laparoscopic cholecystectomy in 200 consecutive patients using an ultrasonically activated scalpel. Surg Laparosc Endosc. 1995 Aug;5(4):255-62. PMID 7551275
- [Result] Rothenberg SS. Laparoscopic splenectomy using the harmonic scalpel. J Laparoendosc Surg. 1996 Mar;6 Suppl 1:S61-3. PMID 8832930
- [Result] Koh YW, Park JH, Lee SW, Choi EC. The harmonic scalpel technique without supplementary ligation in total thyroidectomy with central neck dissection: a prospective randomized study. Ann Surg. 2008 Jun;247(6):945-9. doi: 10.1097/SLA.0b013e31816bcd61. PMID 18520221
- [Result] Markkanen-Leppanen M, Pitkaranta A. Parotidectomy using the Harmonic scalpel. Laryngoscope. 2004 Feb;114(2):381-2. doi: 10.1097/00005537-200402000-00038. No abstract available. PMID 14755223
- [Result] Siperstein AE, Berber E, Morkoyun E. The use of the harmonic scalpel vs conventional knot tying for vessel ligation in thyroid surgery. Arch Surg. 2002 Feb;137(2):137-42. doi: 10.1001/archsurg.137.2.137. PMID 11822946
- [Result] Miccoli P, Materazzi G, Fregoli L, Panicucci E, Kunz-Martinez W, Berti P. Modified lateral neck lymphadenectomy: prospective randomized study comparing harmonic scalpel with clamp-and-tie technique. Otolaryngol Head Neck Surg. 2009 Jan;140(1):61-4. doi: 10.1016/j.otohns.2008.10.003. PMID 19130963
- [Result] Walen SG, Rudmik LR, Dixon E, Matthews TW, Nakoneshny SC, Dort JC. The utility of the harmonic scalpel in selective neck dissection: a prospective, randomized trial. Otolaryngol Head Neck Surg. 2011 Jun;144(6):894-9. doi: 10.1177/0194599811403874. Epub 2011 Mar 31. PMID 21493266
- [Result] Gall AM, Sessions DG, Ogura JH. Complications following surgery for cancer of the larynx and hypopharynx. Cancer. 1977 Feb;39(2):624-31. doi: 10.1002/1097-0142(197702)39:23.0.co;2-7. PMID 837342
- [Result] Yarington CT Jr, Yonkers AJ, Beddoe GM. Radical neck dissection. Mortality and morbidity. Arch Otolaryngol. 1973 Apr;97(4):306-8. doi: 10.1001/archotol.1973.00780010316003. No abstract available. PMID 4699538
- [Result] Hambley R, Hebda PA, Abell E, Cohen BA, Jegasothy BV. Wound healing of skin incisions produced by ultrasonically vibrating knife, scalpel, electrosurgery, and carbon dioxide laser. J Dermatol Surg Oncol. 1988 Nov;14(11):1213-7. doi: 10.1111/j.1524-4725.1988.tb03478.x. PMID 3141490
- [Result] Mantke R, Halangk W, Habermann A, Peters B, Konrad S, Guenther M, Lippert H. Efficacy and safety of 5-mm-diameter bipolar and ultrasonic shears for cutting carotid arteries of the hybrid pig. Surg Endosc. 2011 Feb;25(2):577-85. doi: 10.1007/s00464-010-1224-6. Epub 2010 Jul 8. PMID 20614136
- [Result] Emam TA, Cuschieri A. How safe is high-power ultrasonic dissection? Ann Surg. 2003 Feb;237(2):186-91. doi: 10.1097/01.SLA.0000048454.11276.62. PMID 12560776
- [Result] Fazan VP, da Silva JH, Borges CT, Ribeiro RA, Caetano AG, Filho OA. An anatomical study on the lingual-facial trunk. Surg Radiol Anat. 2009 Apr;31(4):267-70. doi: 10.1007/s00276-008-0439-x. Epub 2008 Nov 13. PMID 19005610
- [Result] Williams MA, Nicolaides AN. Predicting the normal dimensions of the internal and external carotid arteries from the diameter of the common carotid. Eur J Vasc Surg. 1987 Apr;1(2):91-6. doi: 10.1016/s0950-821x(87)80004-x. PMID 3503020
- [Result] Cappiello J, Piazza C, Giudice M, De Maria G, Nicolai P. Shoulder disability after different selective neck dissections (levels II-IV versus levels II-V): a comparative study. Laryngoscope. 2005 Feb;115(2):259-63. doi: 10.1097/01.mlg.0000154729.31281.da. PMID 15689746
- [Result] Erisen L, Basel B, Irdesel J, Zarifoglu M, Coskun H, Basut O, Tezel I, Hizalan I, Onart S. Shoulder function after accessory nerve-sparing neck dissections. Head Neck. 2004 Nov;26(11):967-71. doi: 10.1002/hed.20095. PMID 15459926
- [Result] El Ghani F, Van Den Brekel MW, De Goede CJ, Kuik J, Leemans CR, Smeele LE. Shoulder function and patient well-being after various types of neck dissections. Clin Otolaryngol Allied Sci. 2002 Oct;27(5):403-8. doi: 10.1046/j.1365-2273.2002.00604.x. PMID 12383306
- [Result] Celik B, Coskun H, Kumas FF, Irdesel J, Zarifoglu M, Erisen L, Onart S. Accessory nerve function after level 2b-preserving selective neck dissection. Head Neck. 2009 Nov;31(11):1496-501. doi: 10.1002/hed.21112. PMID 19399751
- [Derived] Shin YS, Koh YW, Kim SH, Choi EC. The efficacy of the harmonic scalpel in neck dissection: a prospective randomized study. Laryngoscope. 2013 Apr;123(4):904-9. doi: 10.1002/lary.23704. Epub 2012 Dec 3. PMID 23208767